CLINICAL TRIAL: NCT05254314
Title: Glucagon-Like Peptide-1 Receptor Agonist Treatment in Adult, Obesity-related, Symptomatic Asthma (GATA-3)
Brief Title: Glucagon-Like Peptide-1 Receptor Agonist in the Treatment of Adult, Obesity-related, Symptomatic Asthma (GATA-3)
Acronym: GATA-3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Katherine Cahill, MD, Medical Director of Asthma Clinical Research, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT-U01-VAN-003; U01AI155299 (NIH)
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Asthma
Keywords: Asthma; Obesity; Semaglutide; Glucagon-like peptide-1 receptor agonist; www.tnasthmaobesitystudy.com
MeSH Terms: conditions — Asthma; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, placebo-controlled, single-center, proof-of-concept study with 2 treatment arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Drug (Semaglutide) (Experimental): Semaglutide 2.4mg once weekly
  Interventions: Drug: Semaglutide Pen Injector 2.4mg weekly
- Placebo (Placebo Comparator): Placebo 2.4mg once weekly
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Semaglutide Pen Injector 2.4mg weekly — Once weekly subcutaneous injection
  Other Names: Wegovy
  Arms: Study Drug (Semaglutide)
Other: Placebo — Once weekly subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a randomized placebo-controlled trial of semaglutide, an FDA-approved therapy for the treatment of type 2 diabetes mellitus and obesity, in adults with symptomatic asthma despite the use of inhaled steroids and with excess body weight. This study will test the central hypothesis that semaglutide will improve asthma control and reduce airway inflammation due to direct effects on the respiratory tract in adult asthma associated with obesity.

DETAILED DESCRIPTION:
This is a proof-of-principal randomized, double-blind, placebo-controlled, single-site clinical trial of semaglutide in adult (age 18 or older, n=100), obesity-related (BMI≥30), symptomatic asthma without type II diabetes. This study will monitor clinical asthma symptom and quality of life questionnaires and airway function to determine the effect of semaglutide on asthma control. Markers of respiratory tract and adipose tissue inflammation will be monitored to determine the effect of semaglutide on airway inflammation. Study participants will be monitored for 4 weeks before assignment to treatment with the study drug for 24 weeks followed by a 2 week final monitoring period.

ELIGIBILITY:
Inclusion Criteria:

1. . Subject must be able to understand and provide informed consent.
2. Males and females age 18 or older
3. Obesity defined as body mass index (BMI) >=30, or >=27 in the setting of >=1 weight-related comorbidity:

   * clinically documented hypertension (>130 mmHg systolic or >85 mmHg diastolic or treatment) in the prior year or during run-in
   * clinically documented dyslipidemia (Triglycerides ш 150 mg/dl, HDL <40 mg/dl in males or <50 mg/dl in females, >=130 mg/dl or treatment) in the prior year or during run-in
   * current obstructive sleep apnea treatment
   * documented pre-diabetes defined by A1c 5.7-<6.5 in the prior year or during run-in
   * clinically documented cardiovascular disease
4. History of physician-diagnosed asthma
5. Persistent Asthma as determined by the requirement of at least medium-dose daily inhaled corticosteroid or more
6. Symptomatic asthma with an ACQ-6 score >=1.5 at enrollment and at the time of randomization
7. Patient report of stable asthma controller regimen for the prior 8 weeks
8. Evidence of bronchodilator responsiveness (>=12% and at least 200 mL increase in FEV1) or airway hyperresponsiveness with a Methacholine PC20 <=16 mg/mL or PD20 <=400 mcg in the prior year
9. Female subjects of childbearing potential must have a negative pregnancy test upon study entry
10. Female subjects of childbearing potential must agree to use a highly effective birth control method (e.g. hormonal, surgical or abstinence) for the duration of the study

Exclusion Criteria:

At enrollment:

1. Inability or unwillingness of a subject to give written informed consent or comply with the study protocol
2. Diagnosis of type I or type II diabetes mellitus (DM) or HbA1c ≥6.5 on screening labs
3. Use of >8 puffs/inhalations of short-acting bronchodilators most days in the previous week (i.e. answer to question #6 on ACQ-6 = 4, 5, or 6)
4. Oxygen saturation < 94% on room air
5. Patient-reported Tobacco, e-cigarette, or smoked marijuana use within 12 months#, or >10 pack-years of use*

   * Can still be enrolled if ≥40 years old, smoked <20 pack years, none within 12 months#, and demonstrate a post-bronchodilator FEV1/FVC ratio of >0.7 or a DLCO z-score of -1.645 or greater (or the equivalent ≥ 75% of predicted) documented in prior 12 months or during run-in

     * Smoking equivalent pack years. One pack of cigarettes a day for 1 year is equivalent to:
   * 1 cigar or pipe per day for 1 year
   * Smoked hookah or shisha =1 session per day for 1 year
   * Vaped e-cigarettes =0.5 mLs e-liquid per day for 1 year, or =1 cartridge/tank/pod per day for 1 year
   * 1 use of inhaled marijuana per day for 1 year

     #Use of any inhalant >1 time weekly in the past year is considered use within 12 months.
   * Active smoking of conventional tobacco, inhaling of marijuana or other drugs, or vaping of e-cigarettes or vape pods >1 time per week in the past year.
   * Any form of tobacco qualifies, such as: 1 cigarette, 1 hookah or shisha sessions, 1 cigar, 1 pipe, etc.
   * Any electronic (e)-device included: e-cigarette e-cig, mod, vape pen, JUUL, e-cigar, e-hookah, e-pipe, vape pods, etc.
   * Any form of inhaled marijuana, including smoking marijuana leaves or inhaling THC via e-cigarette or device
6. Pregnancy by urine testing, current lactation, or plans to become pregnant during the study period
7. Pharmaceutical weight loss treatment for >7 days in the prior 90 days at enrollment
8. Previous surgical weight loss treatment. Can still be enrolled if surgery > 5 years ago and evidence of stable or increasing weight in the prior 3-12 months.
9. Personal history of pancreatitis as determined by history
10. Personal or family history of medullary thyroid cancer by history or multiple endocrine neoplasia syndrome type 2
11. Personal history of gallstone disease without previous cholecystectomy
12. Personal history of gastroparesis
13. Personal history of hypersensitivity to semaglutide
14. Personal history of hypersensitivity to local amide type (ex. Lidocaine) anesthetics
15. Use of antidiabetic agent, other than metformin, including GLP-1R agonist in the previous 90 days. Metformin is allowed provided the dose has been stable in the 90 days prior to screening and will remain stable for the duration of the trial.
16. Use of systemic glucocorticoids in the past 28 days
17. Use of monoclonal antibody for the treatment of asthma in the past 120 days
18. Myocardial infarction, unstable angina, stroke, or heart failure (NYHA class II) within 1 year by history
19. Patient report and confirmed by review of historical diagnostic testing by study physician of other physician-diagnosed chronic respiratory diseases: COPD, cystic fibrosis, pulmonary hypertension, interstitial lung disease, sarcoidosis, bronchiectasis
20. History of physician-diagnosed immune deficiency.
21. History of physician-diagnosed malignancy (other than excised non-melanoma skin cancer) in the past 5 years.
22. Current uncontrolled hypertension (systolic >150, diastolic >90) or untreated hyperthyroidism
23. Current, diagnosed or self-reported drug or alcohol abuse that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements.
24. Use of investigational drugs within 20 weeks of participation, other than vaccines and/or treatments for SARS-CoV-2 authorized for emergency use
25. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the subject's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

    At randomization:
26. Screening creatinine elevation with EGFR<30 ml/min/1.73 m2 collected at visit 1a
27. Compliance to baseline asthma inhaler therapy of <80% during run-in, at the time of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The efficacy of semaglutide on asthma control questionnaire-7 score in subjects with symptoms, persistent asthma and obesity. | Baseline to week 12
  The primary clinical outcome is the difference between the treatment and placebo groups in change from baseline in asthma control questionnaire (ACQ)-7 score to week 12. The ACQ-7 scale ranges from 0-6 with lower scores indicating better asthma control.
The impact of semaglutide once weekly on serum periostin in subjects with symptomatic, persistent asthma and obesity. | Baseline to week 4
  The primary mechanistic outcome is the difference between the treatment and placebo groups in change from baseline in serum periostin at week 4.

SECONDARY OUTCOMES:
The impact of semaglutide on weight loss over time. | Baseline to week 24
  The change from baseline in weight to week 24.
The efficacy of semaglutide once weekly on asthma control questionnaire-6 score in subjects with symptomatic, persistent asthma and obesity | Baseline to week 12
  The change from baseline in ACQ-6 score to week 12. The ACQ-6 scale ranges from 0-6 with lower scores indicating better asthma control.
The maximal dose of semaglutide tolerated in persistent asthma with obesity. | Baseline to week 24
  The maximum tolerated dose of the investigational product at week 24.
Incidence of treatment-emergent adverse events from semaglutide in persistent asthma with obesity. | Baseline to week 26
  The treatment-emergent adverse events from first dose to the completion of follow up at week 26.
The change in exhaled nitric oxide from semaglutide to week 12. | Baseline to week 4 and week 12
  The change from baseline in exhaled nitric oxide at weeks 4 and 12.
The change in serum periostin from semaglutide to week 12. | Baseline to week 4 and week 12
  The change from baseline in serum periostin at week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Cahill, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Tomasello A, Bacharier LB, Becker PM, Dempsey C, Wu P, Peebles RS, Niswender K, Dupont WD, Bernard G, Cahill KN. Untangling obese asthma: Design of proof-of-concept study of semaglutide in poorly controlled asthma. J Allergy Clin Immunol Glob. 2025 Dec 17;5(2):100627. doi: 10.1016/j.jacig.2025.100627. eCollection 2026 Mar. PMID 41567689
- See also: Study Approved Website — https://www.tnasthmaobesitystudy.com/